CLINICAL TRIAL: NCT05136482
Title: Use of a Continuous Cold-flow Cryocompression Device to Reduce the Skin Temperature of the Knee to the Therapeutic Range of 10-15℃: a Randomised Controlled Trial
Brief Title: Skin Temperature Changes When Using a Cryocompression Device
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Winchester (Other)
Collaborators: Physiolab Technologies Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: HWB_REC_210927_Faulkner
Record Dates: First submitted 2021-11-04; First posted 2021-11-29 (Actual); Last update posted 2022-05-19 (Actual); Status verified 2022-05

CONDITIONS: Temperature Change, Body
MeSH Terms: conditions — Body Temperature Changes

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Control (No Intervention): Participants will wear the cryocompression device for 30 mins without any cold or pressure being applied to the lower limb by the cuff.
- Condition A (Experimental): Participants will wear the cryocompression device for 30 minutes while ice-water at a temperature of 6℃ and a pressure of 25 mmHg is applied to the lower limb by the cuff.
  Interventions: Device: Cryocompression
- Condition B (Experimental): Participants will wear the cryocompression device for 30 minutes while ice-water at a temperature of 8℃ and a pressure of 25 mmHg is applied to the lower limb by the cuff.
  Interventions: Device: Cryocompression
- Condition C (Experimental): Participants will wear the cryocompression device for 30 minutes while ice-water at a temperature of 10℃ and a pressure of 25 mmHg is applied to the lower limb by the cuff.
  Interventions: Device: Cryocompression
- Condition D (Experimental): Participants will wear the cryocompression device for 30 minutes while ice-water at a temperature of 12℃ and a pressure of 25 mmHg is applied to the lower limb by the cuff.
  Interventions: Device: Cryocompression

INTERVENTIONS:
Device: Cryocompression — A cryocompression device will be attached to the lower limb of participants using a cuff spanning from the mid-thigh to mid-calf. The device will exert a constant pressure of 25 mmHg throughout each test session. The device will pump temperature-controlled cold water through the cuff in order to reduce the skin temperature around the knee (and intra-articular temperature). Depending on the condition, the temperature of the water being pumped through the device will be either 6, 8, 10, or 12℃. Each test session will last for 30 minutes. Participants will take part in all conditions, with at least 24 hours rest in between test sessions. Skin temperature around the knee will be measured prior to the cryocompression device being applied; every 5 minutes during the 30 minute test; and every 5 minutes after the test until skin temperature >15℃.
  Arms: Condition A; Condition B; Condition C; Condition D

SUMMARY:
Cryotherapy after surgery is widely utilised and has numerous practical applications for post-operative rehabilitation. Previous research has suggested that during cold therapy, the skin temperature of the knee should be reduced to 10-15°C to maximise the therapeutic benefits of cooling while avoiding the risk of cold injuries such as nerve damage and frostbite (Wilke and Weiner, 2003; Bleakley, McDonough and MacAuley, 2004). The temperature range at which a device cryocompression device should be set in order to achieve a skin temperature within the therapeutic range of 10-15°C is unknown. Furthermore, there is evidence to suggest that the temperature of the device does not equal that to which the skin is reduced, plus different devices do not achieve the same reduction in skin temperature despite the ice-water within the knee sleeve being maintained at similar temperatures (Selfe et al., 2009). Therefore, it is not sufficient to assume that the temperature setting of a cryo-compression device reflects the skin temperature achieved.

The aim of this study is to determine which temperature of ice-water flowing through a Physiolab S1 cryocompression device is able to reduce skin temperature around the knee to within the previously stated therapeutic range.

DETAILED DESCRIPTION:
Design This prospective randomised controlled trial will recruit healthy adult volunteers from a university population to participate. Each participant will take part in each condition within the study in order to eliminate the risk of demographic factors confounding the results: Conditions will be conducted in a random order and will be named: control, A, B, C, and D. The control condition will involve the cryocompression device being worn without any ice-water being circulated through the knee sleeve. Conditions A, B, C, and D will involve the device being worn while ice-water is circulated through the knee sleeve at a maintained temperature of 6°C, 8°C, 10°C, or 12°C, respectively. Randomisation will be performed using a computer random number generator.

Protocol All eligible participants will first be required to provide informed consent prior to their participation in the study. Once this has been obtained, participants will each attend a single testing session that should last no longer than 60 minutes. The height and mass of the participants will first be measured in order to calculate BMI, and participants' age and sex will be recorded to allow for later analysis to determine any confounding influence of these factors on the results.

Participants will be required to remain in a seated position with their leg in full extension and elevated, parallel to the floor, for the duration of each test session. The leg that will be used for the study will be randomly selected for each participant, and will remain the same for each condition. A k-type thermocouple will be taped 20 mm distal to the patella and the Physiolab S1 cryocompression device will then be attached to the leg of the participant. Depending on the condition to which a participant has been assigned for a given test, the S1 will maintain the temperature of the water flowing through the device at either 6, 8, 10, or 12℃. The control condition will involve the device being applied to the leg with no ice/water flowing through the cuff. The cuff will be worn for 30 minutes as per the manufacturers guidelines for cold therapy treatments. After 30 minutes, the cuff will be removed. If the temperature of the skin has been reduced to within 10-15℃, skin temperature will continue to be monitored every 5 minutes after the cuff has been removed until it rises above 15℃, at which point the test will end. If the skin temperature is not reduced to within 10-15℃ while the cuff is worn, then the test will end after the cuff is removed at 30 minutes. Upon completion of the test, the temperature sensor will be removed from the leg of the participant; thus completing their participation in the test.

Analysis The data will be analysed to detect any differences during testing compared to baseline measures, and between groups. All data will be first subjected to a Kolmogorov-Smirnov test to assess whether they are normally distributed. A repeated measures analysis of variance will be performed on all normally distributed data. A Friedman test will be performed on any data that are not normally distributed.

Ethical issues There is a low risk of cold injury to participants if their skin temperature reduces to <10℃. Skin temperature will be monitored every 5 minutes throughout the study and testing will be terminated if a participant's skin temperature dips below this threshold. Therefore, the risk to participants in this study is minimal.

Participants have the right to withdraw themselves and any collected data from the study at any time during and after their participation, without having to give a reason. They also have the right to terminate a test session at any time. Testing shall also be terminated as a result of any adverse reactions that emerge. Adverse reactions (e.g. pain) to the testing protocol are not expected due to the low-risk nature of the study, however any that occur shall be recorded and monitored until things return to baseline/normal. In order to monitor any pain/discomfort that might occur, a Visual Analogue Scale (0-10 scale) will be within sight of the participant at all times during testing: a test will be terminated if reported pain/discomfort exceeds 5/10, though none is expected. Any reported pain (or other adverse reactions) shall be stored along with the data collected for that participant. If a test is terminated for a reason that could be mitigated in future, participants will be offered the opportunity to repeat the test another day, should they wish to continue taking part in the study. If a test is terminated due to an adverse reaction that can not be mitigated in future, the participant (and any collected data) will be thanked for their time and withdrawn from the study.

ELIGIBILITY:
Inclusion Criteria:

* >18 years of age.

Exclusion Criteria:

* BMI >40 kg/m2

  * History of nerve damage or sensory deficit in the lower limbs (including frostbite)
  * Hypersensitivity to cold, including hives
  * Active inflammation or pain of the knee
  * History of thrombosis, embolism, or other conditions related to impaired peripheral circulation
  * Suffering from diagnosed diabetes, multiple sclerosis, rheumatoid arthritis, spinal cord injury, cardio-vascular disease, hypertension, Raynaud disease, cryoglobulinemia, or haemoglobinuria
  * Confirmed or suspected tissue infection, an unstable fracture, a skin condition, or a tumour in the treatment area
  * Cognitive impairment or communication barriers

These criteria have been selected in accordance with the common contraindications for cold therapy (Selfe et al, 2009; Fang et al, 2012; Waterman et al, 2012) and those laid out in the manufacturer's guidelines of the specific device to be used (S1; Physiolab Technologies Ltd)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2021-11-10 (Actual); Primary Completion 2022-05-11 (Actual); Study Completion 2022-05-11 (Actual)

PRIMARY OUTCOMES:
Skin Temperature | up to 14 days
  Skin temperature will be measured using a thermocouple positioned 20 mm distal to the patella. This sensor will be attached prior to the cryocompression device being applied, and will remain in place until the testing session is complete and skin temperature is >15℃. (The therapeutic skin temperature range for cryotherapy is thought to be 10-15℃). Temperature will be measured prior to the cryocompression device being applied; every 5 minutes during the test; and every 5 minutes after a test until the skin temperature reaches >15℃.

CONTACTS AND LOCATIONS:
Overall Officials: James Faulkner, PhD, Principal Investigator — University of Winchester
Locations (1):
- Physiology Laboratory, Winchester, United Kingdom

IPD SHARING:
Plan to Share IPD: No
No individual data will be shared outside of the researchers directly involved in the data collection itself.

REFERENCES:
- [Background] Wilke B, Weiner RD. Postoperative cryotherapy: risks versus benefits of continuous-flow cryotherapy units. Clin Podiatr Med Surg. 2003 Apr;20(2):307-22. doi: 10.1016/S0891-8422(03)00009-0. PMID 12776983
- [Background] Bleakley C, McDonough S, MacAuley D. The use of ice in the treatment of acute soft-tissue injury: a systematic review of randomized controlled trials. Am J Sports Med. 2004 Jan-Feb;32(1):251-61. doi: 10.1177/0363546503260757. PMID 14754753
- [Background] Selfe J, Hardaker N, Whittaker J and Hayes C. An investigation into the effect on skin surface temperature of three cryotherapy modalities. Thermology International. 2009; 19(4): 121-126.
- [Background] Fang L, Hung CH, Wu SL, Fang SH, Stocker J. The effects of cryotherapy in relieving postarthroscopy pain. J Clin Nurs. 2012 Mar;21(5-6):636-43. doi: 10.1111/j.1365-2702.2010.03531.x. Epub 2011 Feb 20. PMID 21332855
- [Background] Waterman B, Walker JJ, Swaims C, Shortt M, Todd MS, Machen SM, Owens BD. The efficacy of combined cryotherapy and compression compared with cryotherapy alone following anterior cruciate ligament reconstruction. J Knee Surg. 2012 May;25(2):155-60. doi: 10.1055/s-0031-1299650. PMID 22928433